CLINICAL TRIAL: NCT03809819
Title: Urogynecological and Sexual Functions After Laparoscopic Vecchietti Vaginoplasty
Brief Title: Urogynecological and Sexual Functions After Vecchietti Operation
Status: Completed | Type: Observational
Sponsor: Medical University of Lublin (Other)
Responsible Party: Principal Investigator, Paweł Miotła, Clinical Professor, Medical University of Lublin
Other Study IDs: 03/2019
Record Dates: First submitted 2019-01-16; First posted 2019-01-18 (Actual); Last update posted 2019-01-18 (Actual); Status verified 2019-01

CONDITIONS: Mayer-Rokitansky-Kuster Syndrome
Keywords: Laparoscopic Vecchietti vaginoplasty; sexual function; urinary incontinence
MeSH Terms: conditions — Mullerian aplasia; Urinary Incontinence

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients with MRKHS: Thirteen patients with MRKHS who underwent laparoscopic Vecchietti vaginoplasty
  Interventions: Procedure: laparoscopic Vecchietti vaginoplasty; Diagnostic Test: FSFI questionnaire; Diagnostic Test: UDI-6 questionnaire; Diagnostic Test: IIQ-7 questionnaire
- Control group: A control group of 13 age-matched, childless, sexually active women
  Interventions: Diagnostic Test: FSFI questionnaire; Diagnostic Test: UDI-6 questionnaire; Diagnostic Test: IIQ-7 questionnaire

INTERVENTIONS:
Procedure: laparoscopic Vecchietti vaginoplasty — Patients who underwent laparoscopic Vecchietti vaginoplasty
  Groups: Patients with MRKHS
Diagnostic Test: FSFI questionnaire — Completion of FSFI questionnaire
Diagnostic Test: UDI-6 questionnaire — Completion of UDI-6 questionnaire
Diagnostic Test: IIQ-7 questionnaire — Completion of IIQ-7 questionnaire

SUMMARY:
The aim of this study was to establish the urogynecological and sexual functions after Vecchietti operation.

DETAILED DESCRIPTION:
Thirteen patients with MRKHS who underwent laparoscopic Vecchietti vaginoplasty were included. A control group of 13 age-matched, childless, sexually active women were examined during the same period. All patients underwent the basic evaluation of anatomical outcomes. Sexual outcomes were established by polish validated FSFI questionnaire. Continence status was assessed by polish validated UDI-6 and IIQ-7 questionnaires. The UDI-6 is subdivided in three domains: stress incontinence, irritative and obstructive discomfort. The IIQ-7 measures the implications of urinary incontinence for normal daily functioning.

ELIGIBILITY:
Inclusion Criteria:

* patients with MRKHS who underwent laparoscopic Vecchietti vaginoplasty
* control group of 13 age-matched, childless, sexually active women

Exclusion Criteria:

* unability to understand informed consent

Age Groups: Child, Adult, Older Adult
Study Population: Thirteen patients with MRKHS who underwent laparoscopic Vecchietti vaginoplasty were included. A control group of 13 age-matched, childless, sexually active women were examined during the same period
Sampling Method: Probability Sample
Enrollment: 26 (Actual)
Dates: Start 2011-01-01 (Actual); Primary Completion 2018-12-31 (Actual); Study Completion 2018-12-31 (Actual)

PRIMARY OUTCOMES:
sexual functions after Vecchietti operation | 8 years
  assessment of sexual functions after Vecchietti operation with the use of The Female Sexual Function Index (FSFI) questionnaire
Urinary incontinence after Vecchietti operation | 8 years
  assessment of Urinary incontinence after Vecchietti operation with the use of the Urinary Distress Inventory (UDI 6) and the Incontinence Impact Questionnaire (IIQ 7)

CONTACTS AND LOCATIONS:
Overall Officials: Paweł Miotła, PhD, Principal Investigator — Medical University in Lublin

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Adamiak-Godlewska A, Skorupska K, Rechberger T, Romanek-Piva K, Miotla P. Urogynecological and Sexual Functions after Vecchietti Reconstructive Surgery. Biomed Res Int. 2019 Feb 25;2019:2360185. doi: 10.1155/2019/2360185. eCollection 2019. PMID 30931323